CLINICAL TRIAL: NCT05700383
Title: The Thrive Study: Improving Multimodal Physical Function in Adults With Heterogenous Chronic Pain: Multi-site Feasibility RCT
Brief Title: The Thrive Study: Improving Multimodal Physical Function in Adults With Heterogenous Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Rush University Medical Center (Other); Duke University (Other); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Ana-Maria Vranceanu, PhD, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023P000321; 1R01AT012069-01 (NIH)
Record Dates: First submitted 2023-01-17; First posted 2023-01-26 (Actual); Results first posted 2025-07-16 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Chronic Pain
Keywords: Chronic Pain; Physical Function; Mindfulness
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GetActive-Fitbit (Experimental): GetActive-Fitbit is an adaptation of the original GetActive-Fitbit program, a mind-body program for the unique needs of individuals with chronic musculoskeletal pain that incorporates activity skills to help individuals improve all aspects of physical function. The GetActive-Fitbit sessions address mind-body skills (e.g., mindfulness, deep breathing, self-compassion), walking skills (e.g., step goals, quota-based pacing), and skills to change thinking (e.g., identify unhelpful thoughts about pain and activity, challenging thoughts). The format is a 10-week program delivered in-person with weekly group sessions and home practice of skills and walking.
  Interventions: Behavioral: GetActive-Fitbit
- Healthy Living for Pain (Active Comparator): Healthy Living for Pain is an active intervention that will be dose, attention, and time matches to the GetActive-Fitbit program. Healthy Living for Pain is an adaptation of the Health Enhancement Program, developed by Dr. Vranceanu and colleagues from Stony Brook, with adjustments for patients with chronic musculoskeletal pain. The Healthy Living for Pain sessions provide educational information on chronic musculoskeletal pain, the role of sleep and nutrition, physical activity, healthcare management, medication use, and social connection. The format is a 10-week program delivered in-person with weekly group sessions and home practice journaling.
  Interventions: Behavioral: Healthy Living for Pain

INTERVENTIONS:
Behavioral: GetActive-Fitbit — GetActive-Fitbit is an adaptation of the original GetActive-Fitbit program, a mind-body program for the unique needs of individuals with chronic musculoskeletal pain that incorporates activity skills to help individuals improve all aspects of physical function. The GetActive-Fitbit sessions address mind-body skills (e.g., mindfulness, deep breathing, self-compassion), walking skills (e.g., step goals, quota-based pacing), and skills to change thinking (e.g., identify unhelpful thoughts about pain and activity, challenging thoughts). The format is a 10-week program delivered in-person with weekly group sessions and home practice of skills and walking.
  Arms: GetActive-Fitbit
Behavioral: Healthy Living for Pain — Healthy Living for Pain is an active intervention that will be dose, attention, and time matches to the GetActive-Fitbit program. Healthy Living for Pain is an adaptation of the Health Enhancement Program, developed by Dr. Vranceanu and colleagues from Stony Brook, with adjustments for patients with chronic musculoskeletal pain. The Healthy Living for Pain sessions provide educational information on chronic musculoskeletal pain, the role of sleep and nutrition, physical activity, healthcare management, medication use, and social connection. The format is a 10-week program delivered in-person with weekly group sessions and home practice journaling.
  Arms: Healthy Living for Pain

SUMMARY:
The investigators aim to conduct a randomized controlled trial to test the feasibility of a mind-body walking program compared to a health education program for individuals with chronic musculoskeletal pain. The investigators will assess the feasibility of recruitment procedures (enrollment, recruitment of racial and ethnic minorities) and intervention delivery (fidelity, adherence, credibility, satisfaction, optimization), following pre-specified benchmarks. Both programs will be delivered in-person.

DETAILED DESCRIPTION:
The investigators aim to conduct a randomized controlled trial to test the feasibility of a mind-body walking program (GetActive-Fitbit) compared to a health education program (Healthy Living for Pain) for individuals with chronic musculoskeletal pain. The investigators will assess the feasibility of recruitment procedures (enrollment, recruitment of racial and ethnic minorities) and intervention delivery (fidelity, adherence, credibility, satisfaction, optimization), following pre-specified benchmarks. Both programs will be delivered in-person.

Each program will consist of ten 60-minute sessions in-person. Participants will receive a treatment manual and ActiGraph watch to assess physical function. There are 3 assessment points consisting of self-report surveys and performance-based measures: baseline, post-program, and 6-month follow-up. All participants will receive access to the other program's manual and website after completing the six-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female outpatients, age 18 years or older
2. Fluent in English
3. Have nonmalignant chronic musculoskeletal pain for more than 3 months
4. Able to perform a 6-minute walk test (6MWT)
5. Owns a smartphone with Bluetooth 4.0 or computer
6. Willingness and ability to participate in one of the 2 programs and to comply with the requirements of the study protocol.
7. Free of concurrent psychotropic medication for at least 2 weeks prior to initiation of treatment, OR stable on current medication for a minimum of 6 weeks and willing to maintain a stable dose
8. Low-level of activity (must meet 2/3 criteria; if difficult to assess, recruiter may ask participant to report their recent step data from their smartphone to better understand their activity level)

   1. Sitting for more than 8 hours/day per self-report
   2. Exercising for fewer than 3 days/week (30+min of exercise constitutes an "exercise day") per self-report
   3. Walking for fewer than 7 days/week (30+min of walking constitutes a "walking day") per self-report

Exclusion Criteria:

1. Diagnosed with a medical illness expected to worsen in the next 6 months (e.g., malignancy)
2. Serious mental illness or instability for which hospitalization may be likely in the next 6 months
3. Current active suicidal ideation reported on self-report
4. Untreated and/or unstable schizophrenia, bipolar disorder, or other psychotic disorder
5. Current, active substance abuse or dependence, and current alcohol dependence within the past 6 months
6. Practice of yoga, meditation, guided imagery or other mind body techniques that elicit the RR, once per week for >45 min 3 times/week within the last 3 months or less.
7. Regular use of Fitbit DMD in the last 3 months
8. Unable to walk/in a wheelchair
9. Mild cognitive decline for participants 65+ only (Short Portable Mental Status Questionnaire; PMSQ 4 or more errors).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ana-Maria Vranceanu, PhD, Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (3):
  - Rush Medical Center, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Duke University, Durham, North Carolina

REFERENCES:
- [Derived] Greenberg J, Hooker JE, McDermott KA, La Camera DE, Brewer JR, Szapary CL, Somers TJ, Keefe F, Kelleher SA, Fisher HM, Burns J, Jeddi R, Kulich R, Polykoff GI, Parker RA, Vranceanu AM; THRIVE Study Team; Diachina A, Hogan S, Chou N, Yates L. Feasibility of a Mind-Body Program for Chronic Pain: A Randomized Clinical Trial. JAMA Netw Open. 2025 Jun 2;8(6):e2515685. doi: 10.1001/jamanetworkopen.2025.15685. PMID 40522662
- [Derived] Hooker JE, Brewer JR, McDermott KA, Kanaya M, Somers TJ, Keefe F, Kelleher S, Fisher HM, Burns J, Jeddi RW, Kulich R, Polykoff G, Parker RA; THRIVE Study Team; Greenberg J, Vranceanu AM. Improving multimodal physical function in adults with heterogeneous chronic pain; Protocol for a multisite feasibility RCT. Contemp Clin Trials. 2024 Mar;138:107462. doi: 10.1016/j.cct.2024.107462. Epub 2024 Jan 28. PMID 38286223

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | GetActive-Fitbit | Healthy Living for Pain
Started | 47 | 45
Completed | 43 | 40
Not Completed | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GetActive-Fitbit | Healthy Living for Pain | Total
Number analyzed (Participants) | 47 | 45 | 92
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.1 (13.6) | 60.1 (14.8) | 57.5 (14.3)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Man | 10 | 13 | 23
  Woman | 36 | 32 | 68
  Gender identity not listed | 1 | 0 | 1
  Prefer not to say | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 32 | 69
  Male | 10 | 13 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 39 | 38 | 77
  Unknown or Not Reported | 5 | 5 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 21 | 20 | 41
  White | 17 | 20 | 37
  More than one race | 5 | 3 | 8
  Unknown or Not Reported | 3 | 1 | 4
Region of Enrollment [Number; unit: participants]
  United States | 47 | 45 | 92
Education [Count of Participants; unit: Participants]
  Less than high school | 1 | 1 | 2
  Completed high school or GED | 12 | 6 | 18
  Some college/Associates degree | 11 | 17 | 28
  Completed 4 years of college | 15 | 10 | 25
  Graduate/professional degree | 6 | 9 | 15
  Choose Not to Answer | 2 | 2 | 4
Employment [Count of Participants; unit: Participants]
  Employed full-time | 9 | 12 | 21
  Employed part-time | 4 | 3 | 7
  Keeping House/Housemaker | 4 | 1 | 5
  Other | 4 | 5 | 9
  Retired | 14 | 16 | 30
  Unemployed | 8 | 5 | 13
  Choose Not to Answer | 4 | 3 | 7
Income [Count of Participants; unit: Participants]
  Less than $10,000 | 6 | 3 | 9
  $10,000 to less than $15,000 | 5 | 5 | 10
  $15,000 to less than $20,000 | 1 | 1 | 2
  $20,000 to less than $25,000 | 3 | 3 | 6
  $25,000 to less than $35,000 | 3 | 5 | 8
  $35,000 to less than $50,000 | 9 | 3 | 12
  $50,000 to less than $75,000 | 4 | 3 | 7
  $75,000 or more | 9 | 11 | 20
  Choose Not to Answer | 7 | 11 | 18
Marital Status [Count of Participants; unit: Participants]
  Single, never married | 16 | 13 | 29
  Married | 16 | 14 | 30
  Living with significant other | 1 | 2 | 3
  Separated/Divorced | 9 | 7 | 16
  Widowed | 2 | 7 | 9
  Choose Not to Answer | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Recruitment Feasibility (Ability)
Description: Ability to enroll 80% or more of the sedentary chronic pain patients who meet study criteria.
Time Frame: 1 Year
Measure: Count of Participants; unit: Participants
Groups:
- All Participants (GetActive Fitbit and Healthy Living for Pain): Includes all individuals who were eligible to participate (adult with chronic musculoskeletal pain) across all three sites.
Arm/Group | All Participants (GetActive Fitbit and Healthy Living for Pain)
Number analyzed (Participants) | 132
Participants | 92

2. Primary Outcome: Recruitment Feasibility (Timeliness) - Number of Participants Recruited in 1 Year
Description: Timeliness of enrollment; we will recruit a sample of 90 patients across the 3 sites over the course of 1 year. Participants will be considered enrolled upon randomization. Assessed by the number of participants enrolled in the study over the course of 1 year. If number enrolled meets or exceeds goal of 90 participants, the benchmark is considered met.
Time Frame: 1 Year
Population: Arms are combined because benchmark is calculated prior to participant randomization to treatment group
Measure: Count of Participants; unit: Participants
Groups:
- Number of Participants Enrolled in a 1 Year Period: Includes the period from recruitment starting to the final enrollment across all three sites.
Arm/Group | Number of Participants Enrolled in a 1 Year Period
Number analyzed (Participants) | 92
Participants | 92

3. Primary Outcome: Feasibility of Recruitment Racial and Ethnic Minorities
Description: 38% or more of the entire sample will be comprised of racial and ethnic minorities, which is consistent with the current USA demographic distribution.
Time Frame: 1 Year
Measure: Count of Participants; unit: Participants
Groups:
- All Participants (GetActive Fitbit and Healthy Living for Pain): Includes all enrolled patients across the three study sites.
Arm/Group | All Participants (GetActive Fitbit and Healthy Living for Pain)
Number analyzed (Participants) | 92
Participants | 50

4. Primary Outcome: Intervention Feasibility/ Adherence to Sessions
Description: ≥80 chronic pain patients attend ≥7/10 sessions for each program (70%)
Time Frame: Post-Test (10 Weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | GetActive-Fitbit | Healthy Living for Pain
Number analyzed (Participants) | 46 | 45
Participants
  Attended ≥7 out of 10 group or make-up sessions | 44 | 37
  Attended <7 out of 10 group or make-up sessions | 2 | 8

5. Primary Outcome: Credibility and Expectancy Scale - Credibility
Description: ≥80 chronic pain patients with credibility scores higher than the Credibility and Expectancy Scale credibility subscale's mid-point, indicating intervention credibility. Credibility subscale scores range from 3 to 27. Higher scores indicate higher perceived credibility for the program.
Time Frame: Baseline (0 Weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | GetActive-Fitbit | Healthy Living for Pain
Number analyzed (Participants) | 41 | 39
Participants
  scored above the scale midpoint | 41 | 34
  scored below the scale midpoint | 0 | 5

6. Primary Outcome: Client Satisfaction Scale
Description: ≥80 chronic pain patients with satisfaction scores higher than the scale's mid-point, indicating intervention satisfaction.
Time Frame: Post-Test (10 Weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | GetActive-Fitbit | Healthy Living for Pain
Number analyzed (Participants) | 42 | 40
Participants
  scored above the scale midpoint | 41 | 30
  scored below the scale midpoint | 1 | 10

7. Primary Outcome: Retention
Description: ≥80 post-treatment, ≥75% 6 months follow up for self-report, performance based and Actigraph data (this includes valid data for all participants).
Time Frame: Post-test (10 weeks), Follow-up (24 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | GetActive-Fitbit | Healthy Living for Pain
Number analyzed (Participants) | 47 | 45
Participants
  Post-Test: Completed self-report, performance-based, and objective data with valid data | 44 | 39
  Post-Test: Did not complete self-report, performance-based, and objective data with valid data | 3 | 6
  Follow-Up: Completed self-report, performance-based, and objective data with valid data | 41 | 37
  Follow-Up: Did not complete self-report, performance-based, and objective data with valid data | 6 | 8

8. Primary Outcome: Assessment Feasibility
Description: We calculated the proportion of assessment procedures that were administered as intended in the the checklists of the study protocol. The number of assessment procedures that were administered in line with the study's protocol checklists was divided by the total number of assessment procedures. The benchmark was set to 90%, i.e., assessment procedures were deemed feasible if ≥90% of assessment procedures were delivered as specified in the protocol.
Time Frame: 1 Year
Population: There are no arms/groups for this outcome because the benchmark was calculated based on percentage accuracy of assessment study procedures as conducted by staff not participants
Measure: Count of Units; unit: Number of assessment procedures
Units Other Than Participants: Number of assessment procedures
Groups:
- Accuracy of Standardized Protocol Checklists: Adherence to standardized protocol for baseline, post-test, and follow-up assessments on a 0-100% scale.
Arm/Group | Accuracy of Standardized Protocol Checklists
Number analyzed (Participants) | 92
Number analyzed (Number of assessment procedures) | 3427
Number of assessment procedures | 3241

9. Primary Outcome: Credibility and Expectancy Questionnaire - Expectancy
Description: ≥80 chronic pain patients with expectancy scores higher than the subscale's mid-point, indicating intervention expectancy. Expectancy subscale scores range from 3 to 27. Higher scores indicate more belief that treatment will help.
Time Frame: Baseline (0 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | GetActive-Fitbit | Healthy Living for Pain
Number analyzed (Participants) | 42 | 39
Participants
  scored above the scale midpoint | 36 | 26
  scored below the scale midpoint | 6 | 13

10. Secondary Outcome: Pain, Enjoyment of Life and General Activity (PEG-3) Scale
Description: Rate of a participant's pain intensity and related interference in enjoyment of life and general activity, using a 0-10 Likert scale. Scores range from 0-30 with higher scores indicating greater pain and interference.
Time Frame: Baseline (0 Weeks), Post-Test (10 Weeks), Follow-Up (24 Weeks)
Population: The number of participants who completed post-test and follow-up surveys was fewer than baselines because of patients discontinuing participation.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GetActive-Fitbit | Healthy Living for Pain
Number analyzed (Participants) | 46 | 45
score on a scale
  Baseline | 6.36 (2.05) | 6.72 (1.78)
  Post-Test: number analyzed (Participants) | 44 | 41
  Post-Test | 5.05 (2.41) | 5.89 (2.26)
  Follow-Up: number analyzed (Participants) | 43 | 40
  Follow-Up | 4.61 (2.04) | 5.27 (2.52)

11. Secondary Outcome: WHO Disability Assessment Schedule 2.0 (WHODAS)
Description: The WHODAS measures level of functioning in six domains: cognition, mobility, self-care, getting along, life activities, and participation. Each question on the scale is measured 0-4. The score range is 0-100, with higher scores indicating more disability.
Time Frame: Baseline (0 Weeks), Post-Test (10 Weeks), Follow-Up (24 Weeks)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GetActive-Fitbit | Healthy Living for Pain
Number analyzed (Participants) | 44 | 45
score on a scale
  Baseline: number analyzed (Participants) | 42 | 45
  Baseline | 48.79 (22.35) | 44.86 (25.04)
  Post-Test: number analyzed (Participants) | 44 | 36
  Post-Test | 35.21 (19.09) | 39.24 (26.02)
  Follow-Up: number analyzed (Participants) | 41 | 37
  Follow-Up | 34.61 (25.03) | 36.93 (25.57)

12. Secondary Outcome: 6 Minute Walk Test (6MWT)
Description: The 6MWT is a performance-based measure that assesses physical function and endurance.
Time Frame: Baseline (0 Weeks), Post-Test (10 Weeks), Follow-Up (24 Weeks)
Population: The number of participants who completed post-test and follow-up assessments was fewer than baselines because of patients discontinuing participation.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | GetActive-Fitbit | Healthy Living for Pain
Number analyzed (Participants) | 47 | 45
meters
  Baseline | 289.62 (77.61) | 260.28 (76.26)
  Post-Test: number analyzed (Participants) | 44 | 40
  Post-Test | 339.20 (80.32) | 307.37 (80.11)
  Follow-Up: number analyzed (Participants) | 42 | 37
  Follow-Up | 316.71 (77.22) | 299.74 (74.87)

13. Secondary Outcome: ActiGraph GT9X
Description: The ActiGraph GT9X is a step count device that objectively measures function (number of steps).
Time Frame: Baseline (0 Weeks), Post-Test (10 Weeks), Follow-Up (24 Weeks)
Population: The number of participants who received an ActiGraph at post-test and follow-up was fewer than baselines because of patients discontinuing participation.
Measure: Mean (Standard Deviation); unit: Steps
Arm/Group | GetActive-Fitbit | Healthy Living for Pain
Number analyzed (Participants) | 46 | 44
Steps
  Baseline | 2641.43 (1735.57) | 3177.11 (2573.83)
  Post-Test: number analyzed (Participants) | 44 | 40
  Post-Test | 3694.77 (2175.43) | 3032.90 (2668.91)
  Follow-Up: number analyzed (Participants) | 42 | 38
  Follow-Up | 3050.62 (2023.89) | 3290.56 (2496.78)

14. Secondary Outcome: PROMIS Depression v1.08b
Description: The PROMIS depression v1.08b measures negative mood, views of self and cognitions on a 5-point scale. Raw scores are converted into a t-score with a mean of 50 and standard deviation of 10. Higher scores indicate more depressive symptoms.
Time Frame: Baseline (0 Weeks), Post-Test (10 Weeks), Follow-Up (24 Weeks)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GetActive-Fitbit | Healthy Living for Pain
Number analyzed (Participants) | 47 | 45
score on a scale
  Baseline | 54.67 (9.48) | 54 (9.54)
  Post-Test: number analyzed (Participants) | 44 | 42
  Post-Test | 52.81 (8.53) | 52.14 (9.49)
  Follow-Up: number analyzed (Participants) | 43 | 40
  Follow-Up | 52.59 (8.75) | 52.82 (10.60)

15. Secondary Outcome: PROMIS Anxiety v1.08a
Description: The PROMIS anxiety v1.08a measures fear, worry, hyperarousal and somatic symptoms. Each item is rated on a 1-5 point Likert Scale and raw scores are converted to t-scores with a mean of 50 and a standard deviation of 10. Higher scores indicating more anxiety symptoms.
Time Frame: Baseline (0 Weeks), Post-Test (10 Weeks), Follow-Up (24 Weeks)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GetActive-Fitbit | Healthy Living for Pain
Number analyzed (Participants) | 47 | 45
score on a scale
  Baseline | 57.25 (10.49) | 56.24 (10.14)
  Post-Test: number analyzed (Participants) | 44 | 42
  Post-Test | 55.04 (9.84) | 54.69 (9.08)
  Follow-Up: number analyzed (Participants) | 43 | 40
  Follow-Up | 53.67 (9.92) | 53.12 (12.97)

16. Secondary Outcome: Pain Catastrophizing Scale (PCS)
Description: A 13-item questionnaire assessing one's tendency to focus on pain-related thoughts and feel helpless and hopeless due to pain on a scale of 0 to 4. Higher scores indicate higher pain catastrophizing. Scores range from 0 to 52.
Time Frame: Baseline (0 Weeks), Post-Test (10 Weeks), Follow-Up (24 Weeks)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GetActive-Fitbit | Healthy Living for Pain
Number analyzed (Participants) | 47 | 45
score on a scale
  Baseline | 20.47 (11.30) | 19.71 (13.56)
  Post-Test: number analyzed (Participants) | 44 | 41
  Post-Test | 11.70 (9.60) | 16.77 (13.81)
  Follow-Up: number analyzed (Participants) | 43 | 40
  Follow-Up | 12.57 (8.86) | 16.20 (13.63)

17. Secondary Outcome: Tampa Kinesiophobia Scale (TSK)
Description: A 17-item questionnaire that assesses fear avoidance and fear of activity. Higher scores indicate higher kinesiophobia. Scores range from 17 to 68.
Time Frame: Baseline (0 Weeks), Post-Test (10 Weeks), Follow-Up (24 Weeks)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GetActive-Fitbit | Healthy Living for Pain
Number analyzed (Participants) | 47 | 39
score on a scale
  Baseline | 39.98 (5.39) | 40.37 (5.84)
  Post-Test: number analyzed (Participants) | 44 | 38
  Post-Test | 34.88 (6.86) | 40.13 (5.70)
  Follow-Up: number analyzed (Participants) | 43 | 38
  Follow-Up | 34.94 (6.00) | 39.20 (7.52)

18. Secondary Outcome: Measure of Current Status (MOCS)
Description: The MOCS questionnaire assesses ability to engage in a series of healthy coping skills (e.g., relaxation, social support, adaptive thinking). Higher scores indicate a stronger ability to recognize stress and cope, with scores ranging from 10 to 50.
Time Frame: Baseline (0 Weeks), Post-Test (10 Weeks), Follow-Up (24 Weeks)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GetActive-Fitbit | Healthy Living for Pain
Number analyzed (Participants) | 47 | 44
score on a scale
  Baseline | 2.27 (0.60) | 2.27 (0.84)
  Post-Test: number analyzed (Participants) | 44 | 41
  Post-Test | 2.50 (0.68) | 2.37 (0.79)
  Follow-Up: number analyzed (Participants) | 43 | 40
  Follow-Up | 2.51 (0.74) | 2.57 (0.83)

19. Secondary Outcome: Cognitive and Affective Mindfulness Scale (CAMS)
Description: Rate of a participant's broad conceptualization of mindfulness, items range from 1-4. Higher values reflect higher levels of mindfulness. Scores range from 12 to 48.
Time Frame: Baseline (0 Weeks), Post-Test (10 Weeks), Follow-Up (24 Weeks)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GetActive-Fitbit | Healthy Living for Pain
Number analyzed (Participants) | 47 | 45
score on a scale
  Baseline | 32.11 (5.68) | 34.43 (7.98)
  Post-Test: number analyzed (Participants) | 44 | 41
  Post-Test | 34.33 (5.97) | 34.32 (7.52)
  Follow-Up: number analyzed (Participants) | 43 | 40
  Follow-Up | 32.96 (6.42) | 35.46 (6.88)

20. Secondary Outcome: Modified Global Impression of Change (MGIC)
Description: 3-items assessing the extent to which patients perceive the intervention improved functioning and symptoms. Each item is rated on a 1-7 point scale with higher scores indicated greater perceived improvement.
Time Frame: Baseline (0 Weeks), Post-Test (10 Weeks), Follow-Up (24 Weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GetActive-Fitbit | Healthy Living for Pain
Number analyzed (Participants) | 44 | 40
score on a scale
  Global Impressions of Change: Pain Management | 6.20 (0.70) | 5.38 (1.23)
  Global Impressions of Change: Physical Function | 5.93 (0.87) | 5.15 (1.29)
  Global Impressions of Change: Emotional Wellbeing | 6.00 (0.75) | 5.40 (1.32)

ADVERSE EVENTS:
Time Frame: 9 months
Arm/Group | GetActive-Fitbit | Healthy Living for Pain
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/45
Serious Adverse Events (participants affected / at risk) | 6/47 | 1/45
Other Adverse Events (participants affected / at risk) | 11/47 | 16/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GetActive-Fitbit (N=47) | Healthy Living for Pain (N=45)
Active Suicidality (Psychiatric disorders) | 1 | 0 — Report of recent, aborted suicide attempt
Hospitalization for high blood pressure (Blood and lymphatic system disorders) | 1 | 0 — Prolonged hospitalization to manage high blood pressure
Kidney Transplant (Renal and urinary disorders) | 1 | 0 — Received a kidney transplant for chronic kidney disease
Hospitalization for blood clot (Blood and lymphatic system disorders) | 1 | 0 — Loss of consciousness and subsequent hospitalization for blood clot in the lungs
Hospitalization for migraine (General disorders) | 1 | 0 — Hospitalized for severe migraine; received lidocaine shots
Hospitalization for neurological symptoms (Nervous system disorders) | 1 | 0 — Admitted to hospital for stroke-like symptoms
Cerebrovascular accident (Vascular disorders) | 1 | 0
Hospitalization for lumbar surgery (Surgical and medical procedures) | 0 | 1 — Repeated unsuccessful lumbar procedures
Hospitalization after emergency room visit (General disorders) | 0 | 1 — Four ER trips with three subsequent hospitalizations
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GetActive-Fitbit (N=47) | Healthy Living for Pain (N=45)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 | 2 — Irritation on wrist after smart-watch wear
Emergency room visit for pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 2 — ER visit for intense pain that did not result in hospitalization
Emergency room visit for urinary tract infection (Renal and urinary disorders) | 1 | 0
Musculoskeletal pain/injury (Musculoskeletal and connective tissue disorders) | 5 | 2
Kidney injury or infection (Renal and urinary disorders) | 1 | 1
Adverse reaction to medical procedure (Injury, poisoning and procedural complications) | 1 | 1
Toxic Multinodular Goiter (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Distress related to intervention homework (Psychiatric disorders) | 0 | 1
Autoimmune disease diagnosis (Immune system disorders) | 0 | 2
Passive death ideation (Psychiatric disorders) | 0 | 1
Motor vehicle collision (General disorders) | 0 | 2
Severe rectal bleeding (Gastrointestinal disorders) | 0 | 1
Partial psychiatric hospitalization (Psychiatric disorders) | 0 | 1
Fall (General disorders) | 0 | 1
Outpatient procedure (Surgical and medical procedures) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-03-21): https://cdn.clinicaltrials.gov/large-docs/83/NCT05700383/Prot_SAP_000.pdf